CLINICAL TRIAL: NCT07131709
Title: Patient Satisfaction With AI Scribes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Papatoetoe Family Doctors (Unknown); The University of Auckland (Unknown)
Responsible Party: Principal Investigator, Keith J Petrie, Professor, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AH29769
Record Dates: First submitted 2025-08-05; First posted 2025-08-20 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: AI (Artificial Intelligence); Patient Satisfaction With AI in Doctors Consultations
Keywords: AI; Patient Satisfaction; Artificial Intelligence; AI in Primary Care; Patient satisfaction with AI; Doctor Consultations
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AI Summary (Experimental): Participants who are randomised to the 'AI Summary' arm will receive an AI-generated summary of their doctors appointment via email.
  Interventions: Other: AI Generated Summary
- AI Summary + Next Steps Plan (Experimental): Participants who are randomised to the 'AI Summary + Next Steps Plan' arm will receive an AI-generated summary of their doctor's appointment via email, as well as an AI-generated plan for their treatment as per the recommendations of the doctor. This may include actionable steps, such as 'collect prescription from pharmacy'.
  Interventions: Other: AI Generated Summary
- Control (No Intervention): The control arm will receive standard care, where no summary of the appointment is emailed.

INTERVENTIONS:
Other: AI Generated Summary — Summary of the doctor's appointment generated by AI (either with or without the Next Steps Plan, depending on the arm participants are allocated to).
  Arms: AI Summary; AI Summary + Next Steps Plan

SUMMARY:
This randomised control trial study explores patient satisfaction with the use of an artificial intelligence (AI) notetaker in doctor's consultations. This involves an AI notetaker being used during doctor's consultations to summarise the conversation between the GP and patient. Patient participants in this study will complete a pre-appointment demographic questionnaire, and attend their doctor's appointment as usual. After the appointment, they will complete a second questionnaire which asks about their experience and satisfaction with the consult, as well as their thoughts towards AI notetakers.

Participants will then be randomised into three groups. One group will receive standard care (no AI summary emailed to them), the second group will be emailed by their doctor an AI-generated summary of the appointment, and the third group will receive the AI summary + a next steps plan. The next steps plan is generated by AI, and outlines steps they need to take after attending their appointment, based on what was discussed with their doctor.

All participants will be emailed a follow-up questionnaire on day three which is tailored to the intervention they received. This re-assesses patient satisfaction with their appointment and the use of AI, as well as their trust in the AI notetaker. Those who receive an AI summary will be asked about their satisfaction with the summary, and those who received an AI summary + next steps plan will be asked about both the summary and next steps plan.

This study will be the first to explore patient satisfaction with the use of an AI scribe in doctor's consultations, and aims to gain a better understanding of patient's perspectives on AI notetakers in primary care settings.

DETAILED DESCRIPTION:
Artificial intelligence (AI) is increasingly being integrated into primary care throughout various physical health contexts. Many clinicians use human-led AI systems to aid with task simplification and documentation in the form of digital scribes. AI scribes record clinical encounters and use natural language processing to convert speech to text, generating a conversation summary. This serves as an efficient and user-friendly tool that can substitute traditional notetaking methods.

While emerging evidence demonstrates the benefits of automating documentation for physicians, there is a paucity of research evaluating patients' satisfaction with AI being used during one-to-one consultations. Understanding patients' satisfaction with the use of AI in primary care settings is important because it can give insight into their perceived benefits and concerns toward the technology. These perceptions can affect patients' level of engagement and rapport with their healthcare provider, which is particularly important for optimising health outcomes.

Artificial intelligence is being utilised across various healthcare contexts, including detecting, diagnosing, and treating various health condition. Research demonstrates that physicians are largely receptive to AI, with one in four doctors using it regularly in some form and increasingly often. To date, research examining patient views on the use of AI in clinical settings remains limited, particularly with respect to primary care settings. Very little research has been conducted to explore patients' perspectives on AI notetakers being used in primary care settings. Most existing research focuses on physician's views on AI in primary settings, or patient's views on AI in specialised health settings. Existing literature across more specialised settings shows that patients are generally receptive toward AI being used during their care, although there is agreement that it should be used as a tool to support clinicians rather than be used unsupervised. For patients to benefit from AI scribes in primary care, they must first be receptive towards its use. Therefore, this is the first study to examine patients' satisfaction and trust with an AI scribe in doctor's consultations. It is important to research this in order to understand their preferred level of engagement with the technology.

This study will address this gap in the literature by providing experimental research on patient's self-reported satisfaction with AI scribes. This research will incorporate patients with a range of ethnicities, ages (18+) and health conditions/concerns. Researching in a primary care setting will enable our study to capture a range of views on artificial intelligence across varying presenting problems, without limiting participants based on their health condition. This study will help to indicate whether patients are receptive to AI notetakers being used during their appointments or not. Understanding people's satisfaction and trust in AI is important because it may effect their level of engagement with their doctor if they frequently use AI.

Providing patients with an AI summary of their appointment may improve overall appointment satisfaction. This intervention will remind patients what was discussed during the appointment (including what actions they are expected to take next), which may improve health outcomes by helping patients to take action on the doctor's recommendations. This intervention will be particularly beneficial for patients with complex health conditions who have to recall a substantial amount of information about their treatment.

ELIGIBILITY:
Inclusion Criteria:

* This study requires participants to have an appointment with the GP involved in this study. Participants must be 18 years or older, be able to read, write, and understand English, able to provide full and informed consent, have access to a device that connects to the internet, and have an email address.

Exclusion Criteria:

* This study has very few exclusion criteria. The only participants who will be excluded are those under the age of 18, those who do not feel able to complete the questionnaires or participate, those who cannot understand/communicate in English (and therefore cannot provide informed consent), and people who do not have an email to be contacted by. This study will allow patient participants with a large variety of presenting health concerns and conditions to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2025-08-11 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | From the participant's recruitment day (which is also their appointment day) until the follow-up questionnaire administered on day three.
  Self-reported patient satisfaction with the use of AI during doctor's consultations, including their overall satisfaction during the appointment, and their satisfaction with the AI summary after the appointment (treatment groups only), collected via questionnaire.
  Adapted from the Patient Satisfaction Questionnaire-III (long form). 'I had enough time to discussed everything with the doctor' (strongly disagree - agree) 'The doctor listened to my concerns' 'I received enough information about my condition/treatment' 'Overall, how satisfied were you with your recent appointment with your doctor?' (Not at all satisfied - extremely satisfied)

SECONDARY OUTCOMES:
Trust in AI | From initial recruitment (also the day of participant's appointment) through to their follow-up questionnaire on day three.
  Will measure self-reported patient trust in AI note-taking software, such as whether participants thought AI would securely store their patient information. Measured via a questionnaire adapted from the Trust in Automation Scale (TIAS), including:
  * 'I trust that the AI notetaker will keep my information private' (strongly disagree - strongly agree)
  * 'I trust that the AI notetaker will securely store my information' (strongly disagree - strongly agree)
  * 'How credible (trustworthy/believable) was the summary' (not credible at all - extremely credible)
  * 'If you were discussing a sensitive topic with your doctor, how comfortable would you be with artificial intelligence being used to take notes?' (extremely uncomfortable - comfortable)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Petrie, Professor of Health Psychology, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- Papatoetoe Family Doctors, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No